CLINICAL TRIAL: NCT02481167
Title: Evaluation of Meibomian Gland Dysfunction in Chinese Old Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: WZ-ZYY-DRYEYE
Record Dates: First submitted 2015-06-15; First posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Dry Eye
Keywords: Aged; Meibomian Glands; dry eye; Elderly
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- group1: This study was consisted of patients with older than 40 years of age who complained with dry eye.

SUMMARY:
The purpose of this study is to identify age-related changes in chinese meibomian glands that may be associated with meibomian gland dysfunction (MGD).

ELIGIBILITY:
Inclusion Criteria:

* have dry eye symptom
* have meibomian gland dysfunction

Exclusion Criteria:

* diabetes
* history of ocular surgery
* systemic disease or inflammation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was consisted of patients with older than 40 years of age who complained with dry eye. The institutional review board of Wenzhou Medical College approved the study protocol, and all patients provided their informed consent.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-04 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Tear film break-up time | 1 year
  Tear film break-up time (TBUT) was evaluated by placing a single fluorescein strip over the inferior tear meniscus after instilling a drop of normal saline.
Lower tear meniscus | 1 year
  Lower tear meniscus was evaluated by keratography
The morphology of meibomian glands | 1 year
  The morphology of meibomian glands was evaluated by keratography

CONTACTS AND LOCATIONS:
Overall Officials: ZHAO YUNE, MS, Study Chair — Wenzhou Medical University
Locations (1):
- Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Li J, Ma J, Hu M, Yu J, Zhao Y. Assessment of tear film lipid layer thickness in patients with Meibomian gland dysfunction at different ages. BMC Ophthalmol. 2020 Oct 6;20(1):394. doi: 10.1186/s12886-020-01667-8. PMID 33023522
- [Derived] Wu Y, Li J, Hu M, Zhao Y, Lin X, Chen Y, Li L, Zhao YE. Comparison of two intense pulsed light patterns for treating patients with meibomian gland dysfunction. Int Ophthalmol. 2020 Jul;40(7):1695-1705. doi: 10.1007/s10792-020-01337-0. Epub 2020 Mar 21. PMID 32200506